CLINICAL TRIAL: NCT05707364
Title: Feasibility and Efficacy Study for a Pre-visit Lab Protocol for Adult Medicine Physicals
Status: Enrolling by invitation | Type: Observational
Sponsor: Endeavor Health (Other)
Collaborators: American Medical Association (Other)
Responsible Party: Principal Investigator, Nadim Ilbawi, Principal Investigator, Clinical Assistant Professor, Endeavor Health
Other Study IDs: EH22-450
Record Dates: First submitted 2023-01-06; First posted 2023-01-31 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Physical Examination; Diagnostic Tests, Routine; Burnout, Professional
Keywords: Feasibility
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Practices Engaged for Pre-Visit Lab Clinic Workflow: Providers and patients/ at the designated practice sites
  Interventions: Behavioral: Pre-visit Lab Workflow

INTERVENTIONS:
Behavioral: Pre-visit Lab Workflow — 1. Based on buy-in from the providers/staff one or both of the practices below will be introduced into the clinic workflow to order pre-visit labs.
     1. All procedures are within the standard of care, only the order of operations is being changed. After sharing lab results with patient from the most recent routine physical, physician records labs for the next calendar year in EMR.
     2. Prior to appointment, Medical Assistant (MA) will review notes and orders to setup pre-visit labs.
  2. Patient contacted to complete labs prior to the scheduled routine physical.
  3. Resulted labs are triaged based on urgency.
  4. After Visit Summary used to communicate about labs and surveys.

SUMMARY:
This is a research study evaluating the implementation of a clinic workflow to encourage pre-visit laboratory testing, such as blood work. The purpose of this research is to understand provider and patient satisfaction with clinic workflows to support pre-visit laboratory tests (blood work) for annual physical and wellness visits. Providers and staff at participating sites will be approached to fill out an anonymous survey regarding experiences with implementation of the pre-visit laboratory testing workflow. Additional data from NorthShore's Enterprise Data Warehouse (EDW) will be collected to assess the pre-lab test rate before implementation, at 6 months, and 12 months, in addition to provider and staff time efficiencies and patient satisfaction as assessed by surveys.

DETAILED DESCRIPTION:
This is a research study about implementing a clinic workflow to encourage pre-visit laboratory testing, such as blood work. Resulting labs is a critical yet time consuming task for primary care clinicians. Ideal and timely management of both normal and abnormal lab results is best done when the patient and clinician are face to face in an office visit. This allows patients to ask questions and clinicians to most efficiently make recommendations, adjust or start medications, or order follow up testing. There is a notable and measurable time commitment to the in-basket burden of sharing lab results via a patient portal or phone calls, advising or counseling on these results and answering subsequent patient inquiries. Furthermore, in a consumer-centric health system and one in which routine blood tests are ordered for employment/insurance purposes and peace of mind, over-ordering of lab testing and the subsequent associated anxiety of out of range results are both costly to the patient and the health care system. Going "upstream" of the in-basket work associated with lab results requires a workflow that maximizes staff time, emphasizes patient engagement and understanding and most efficiently uses clinician time to guide good patient care.

The aims of this research study include to measure the feasibility of implementing a pre-visit lab testing clinic workflow, which involves clinicians using the electronic medical record (EMR) to indicate preferences that upcoming labs be completed prior to their scheduled physical so that results can be discussed during the office visit, and to study the efficacy of a pre-visit lab workflow as it relates to clinician in-basket time, staff time, patient satisfaction, provider satisfaction, and frequency of patient encounters post visit.

The study has multiple components to test these aims. Approximately 4 sites will be engaged to implement the study workflow for all prospective patients seen at the designated offices. Site physicians and their clinic staff will be invited to attend a Lunch & Learn to discuss the intent to implement pre-visit lab testing and confirm the details of the clinic workflow. Data will be reviewed for progress reports and modifications to the clinical workflow can be made at that time to adjust for implementation barriers.

Longitudinal data from a brief survey will be collected from clinical staff (e.g. providers, practice managers, nurses, medical assistants, etc.) at three time points: prior to study implementation, at 6-months of implementation, and at 1-year of implementation. Practices will act as their own controls with their patients with labs resulted on/post-visit compared to those resulted pre-visit. Data sources will include EDW data, Press-Ganey scores, and physician surveys to assess time burden and satisfaction with workflow.

A secondary study component will involve anonymous patient surveys collected at every annual physical or wellness visit for the duration of the study. Additionally, patient data will be collected from existing sources (EPIC/Clarity, Press-Ganey, Enterprise Data Warehouse, billing, etc.) to assess the effectiveness of the workflow as it relates to patient understanding of their care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older.
* Patients must have had an annual physical/ wellness visit within 30 days of completing the survey.
* Patient/ providers willing to complete the survey.

Exclusion Criteria:

• Participants younger than 18 years of age.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 4 NorthShore Medical Group Primary Care (Family Medicine/ Internal Medicine/ non-specialty) sites will be asked to implement the study workflow for all prospective patients (approximately 30,000 total) seen between 11/1/2022- 11/1/2024 at the designated offices.
Sampling Method: Non-Probability Sample
Enrollment: 301000 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pre-lab test rate | 3 months prior to study implementation and then ongoing to month 24 to calculate monthly proportions
  Count of pre-lab tests completed out of the total number of annual physical/wellness visits to participating providers to participating providers

SECONDARY OUTCOMES:
Change from baseline clinician time spent resulting labs | baseline (prior to study implementation), at 6-months of implementation, and at 1-year of implementation
  Time questions asked in provider questionnaire
Change from baseline provider satisfaction | baseline (prior to study implementation), at 6-months of implementation, and at 1-year of implementation
  Agreement metrics (1= Strongly disagree to 5= Strongly agreed) asked in provider questionnaire. Higher scores indicate a better outcome.
Change from baseline patient satisfaction | baseline, 1 year, and 2 year (i.e. annually at every wellness/ annual physical visit)
  Agreement metrics (1= Strongly disagree to 5= Strongly agreed) asked in provider questionnaire. Higher scores indicate a better outcome.
Change from baseline frequency of patient encounters post visit | 3 months prior to study implementation and then ongoing to month 24 to calculate monthly proportions
  Enterprise Data Warehouse data pull

CONTACTS AND LOCATIONS:
Overall Officials: Nadim Ilbawi, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinsky CA, Sinsky TA, Rajcevich E. Putting Pre-Visit Planning Into Practice. Fam Pract Manag. 2015 Nov-Dec;22(6):34-8. No abstract available. PMID 26761083
- [Background] American Medical Association. 10 steps to pre-visit planning that can produce big savings. Sept 4, 2015. https://www.ama-assn.org/practice-management/sustainability/10-steps-pre-visit-planning-can-producebig-savings